CLINICAL TRIAL: NCT05581901
Title: Perioperative Methadone for Ameliorating Postoperative Pain and Reduction in Postoperative Opioid Consumption in Hip Fracture Patients - Dosage Adjusting Pilot-study
Brief Title: Perioperative Methadone in Hip Fracture Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SHS-An-2-2022
Record Dates: First submitted 2022-09-15; First posted 2022-10-17 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Methadone; Pain, Post Operative; Pain, Postoperative; Analgesics, Opioid
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Methadone (Dose 1) (Experimental): Methadone will be administered intravenously at the beginning of surgery, and will only be administered this one time. The gradual upward titration of Methadone will be managed using adaptive platform design. This way the number of patients in each group will be determined by the adaptive platform algorithm.
  Interventions: Drug: Methadone (Dose1)
- Methadone (Dose 2) (Experimental): Methadone will be administered intravenously at the beginning of surgery, and will only be administered this one time. The gradual upward titration of Methadone will be managed using adaptive platform design. This way the number of patients in each group will be determined by the adaptive platform algorithm.
  Interventions: Drug: Methadone (Dose 2)
- Methadone (Dose 3) (Experimental): Methadone will be administered intravenously at the beginning of surgery, and will only be administered this one time. The gradual upward titration of Methadone will be managed using adaptive platform design. This way the number of patients in each group will be determined by the adaptive platform algorithm.
  Interventions: Drug: Methadone (Dose 3)

INTERVENTIONS:
Drug: Methadone (Dose1) — Dose: 0.10mg/kg
  Other Names: Dose 1
  Arms: Methadone (Dose 1)
Drug: Methadone (Dose 2) — Dose: 0.15mg/kg
  Other Names: Dose 2
  Arms: Methadone (Dose 2)
Drug: Methadone (Dose 3) — Dose 0.20mg/kg
  Other Names: Dose 3
  Arms: Methadone (Dose 3)

SUMMARY:
Postoperative analgesic treatment needs to be improved. Numerous studies suggest that a single dose of Methadone given during surgery significantly ameliorates postoperative pain and reduces postoperative opioid consumption. Perioperative methadone is already used in isolated cases such as patients with chronic pain or patients with high morphine tolerance. However, it is not routinely used in the elderly and fragile, and there is insufficient reliable evidence on this treatment and population. Further investigation is highly relevant and necessary.

DETAILED DESCRIPTION:
A multimodal approach and the use of peripheral nerve blocks have improved the treatment of postoperative pain. However, supplemental opioids are predominantly necessary and often continued for months or years after surgery. In fact, continued use of opioids after surgery is an increasing challenge. Consequently, patients undergoing surgery are at risk of experiencing side effects and developing physical as well as psychological addiction to opioids. The most common opioid-related side effects include obstipation, nausea, itchy skin, dry mouth, vertigo, and sedation. The means to decrease the need for opioids in the postoperative phase are in high demand, and therefore the investigation of perioperative Methadone is highly relevant. Methadone is a lipophilic opioid agonist with a large distribution volume and a very long elimination half-life of 15 - 60 hours. It is also an N-methyl D-aspartate (NMDA) receptor antagonist, which attenuates opioid-induced tolerance and hyperalgesia. Furthermore, Methadone inhibits the reuptake of Serotonin and Noradrenalin, which could positively affect the experience of pain in the postoperative phase. Methadone is mostly excreted through the bile and can, therefore, even be used in patients with reduced kidney function. Methadone's analgesic effects occur only eight minutes after intravenous administration. In most studies, methadone is given perioperatively in dosages of 0.10-0.30 mg/kg and is commenced at the induction of anaesthesia or the initiation of surgery. Studies investigating the optimal dosage and time for administration found that patients receiving methadone after the procedure needed twice as much opioid pain medication on postoperative day one compared to patients receiving methadone at anaesthetic induction. These studies also indicate that using smaller dosages such as 5-10 mg, the analgesic duration is only 3-4 hours, whereas doses of 20 mg or more have a clinical effect closely related to the elimination half-life of 15-60 hours without any increased risk for respiratory depression. The aim of this study is to determine the optimal dose of methadone for a future randomized controlled trial (RCT). The objective is to investigate whether doses greater than 0.10 mg/kg are tolerated with no increased risk to respiratory depression, side effects, or prolonged stay in the post-anaesthesia care units (PACU).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a hip fracture on x-rays (collum femoris fractures, pertrochanteric fractures and subtrochanteric fractures).
* Patients must be able to reliably assess their level of pain using the VRS and be able to ask for supplementary analgesics if needed.
* Patients must understand the information given and be able to read and speak Danish.
* Patients must be able to give informed consent.

Exclusion Criteria:

* Polytrauma (defined as a trauma with one or more absolute indications for surgical intervention).
* Previous allergic reactions or hypersensitivity towards Methadone hydrochloride or Sodium-chloride.
* Health conditions preventing treatment, i.e. chronic obstructive pulmonary disease (Gold classification C+D), history with acute asthma attacks or atopic skin conditions, cor pulmonale, raised intracranial pressure or head injury, Pheochromocytoma, history with paralytic ileus, QT interval prolongation, myasthenia gravis, liver disorders or hypotension.
* Concurrent administration with monoamine oxidase inhibitors or within 2 weeks of suspending treatment with these medicinal products.
* Concurrent administration of sedatives, e.g. Benzodiazepines or related drugs.
* Included in other studies (e.g., SENSE-trial).
* Known cognitive disorders e.g., dementia.
* Current drug addiction e.g., opioid addiction or intravenous addiction.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Respiratory depression | 6 hours after surgery
  Occurrence of a respiratory frequency <10/min and oxygen saturation <94 % despite 4 liters of oxygen/min.
Respiratory depression | 24 hours after surgery
  Occurrence of a respiratory frequency <10/min and oxygen saturation <94 % despite 4 liters of oxygen/min.
Respiratory depression | 72 hours after surgery
  Occurrence of a respiratory frequency <10/min and oxygen saturation <94 % despite 4 liters of oxygen/min.

SECONDARY OUTCOMES:
Length of stay at the post anaesthetic care unit | up to 12 hours after surgery
  Hours
Number of times Naloxone was administered | immediately after the surgery (6, 24, 72 hours)
  Numerical
Postoperative opioid consumption | immediately after the surgery (6, 24, 72 hours)
  mean consumption of rescue medication
Opioid-related side-effects | immediately after the surgery (6, 24 hours)
  Opioid-related side-effects will be registered binomial as nausea and vomiting
Postoperative pain | immediately after the surgery (0, 6, 24, 72 hours)
  Patients will be asked to assess pain intensity at the time of arrival from the post-anaesthesia care unit using the Verbal Rating Scale (VRS) consisting of 6 categories where 0 is no pain and 5 is the highest level of pain (worst outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Schønnemann, Principal Investigator — Hospital of Southern Denmark - Aabenraa
Locations (1):
- Sygehus Soenderjylland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedersen AK, Nygaard KH, Petersen SR, Specht K, Strom T, Moos CM, Skjot-Arkil H, Schonnemann JO. Adjusting perioperative methadone dose for elderly and fragile hip fracture patients (MetaHip-trial) - A statistical analysis plan for an adaptive dose-finding trial. Contemp Clin Trials Commun. 2023 Nov 14;36:101228. doi: 10.1016/j.conctc.2023.101228. eCollection 2023 Dec. PMID 38047142